CLINICAL TRIAL: NCT06070779
Title: The Effect of Neurolinguistic Programming on Labor Pain, Fear, Duration and Maternal Satisfaction
Brief Title: Neurolinguistic Programming on Labor Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aysegul Kilicli (Other)
Responsible Party: Sponsor-Investigator, Aysegul Kilicli, Gaziantep University Health Sciences Institute, Department of Nursing, Department of Obstetrics and Gynaecology Nursing, PhD., University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NLP and labor pain
Record Dates: First submitted 2023-09-18; First posted 2023-10-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neurolinguistic Programming; Labor Pain
Keywords: neuro linguistic programming; Labour pain; Labour fear; Labour satisfaction; Labour duration
MeSH Terms: conditions — Labor Pain | interventions — Neurolinguistic Programming

STUDY DESIGN:
Intervention Model Description: randomised controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- neuro linguistic programming group for primiparous (Experimental): NLP application to the experimental group will be done by the researcher Ayşegül Kılıçlı. The application session will 20 minutes. The application will be started in the active phase of labour when the cervical opening is 4 cm.
  In the neuro linguistic programming (NLP); The system of representation of women in practice will be determined first. Then, with the anchoring technique, negative feelings and thoughts about labour will be tried to be erased from the mind or their severity will be reduced. Then, positive feelings and thoughts will be created instead of the mother's negative feelings and thoughts with belief change strategies. Then, with the swish technique, the mother's positive feelings and thoughts about labour will be made aware of and reinforced.
  Interventions: Other: neuro linguistic programming
- control group for primiparous (No Intervention): The control group will not receive only the neuro-linguistic programming, but all other assessments will be parallel to the experimental group (neuro linguistic programming group for primiparous).
- neuro linguistic programmig group for multiparous (Experimental): NLP application to the experimental group will be done by the researcher Ayşegül Kılıçlı. The application session will 20 minutes. The application will be started in the active phase of labour when the cervical opening is 4 cm.
  In the neuro linguistic programming (NLP); The system of representation of women in practice will be determined first. Then, with the anchoring technique, negative feelings and thoughts about labour will be tried to be erased from the mind or their severity will be reduced. Then, positive feelings and thoughts will be created instead of the mother's negative feelings and thoughts with belief change strategies. Then, with the swish technique, the mother's positive feelings and thoughts about labour will be made aware of and reinforced.
  Interventions: Other: neuro linguistic programming
- control group for multiparous (No Intervention): The control group will not receive only the neuro-linguistic programming, but all other assessments will be parallel to the experimental group (neuro linguistic programming group for muliparous).

INTERVENTIONS:
Other: neuro linguistic programming — neuro linguistic programming
  Arms: neuro linguistic programmig group for multiparous; neuro linguistic programming group for primiparous

SUMMARY:
THE EFFECT OF NEURO LINGUISTIC PROGRAMMING ON LABOUR PAIN, FEAR, DURATION AND MATERNAL SATISFACTION

DETAILED DESCRIPTION:
In this study, it is aimed to determine the effect of neuro linguistic programming on labour pain, fear, duration and maternal satisfaction.

Sample size:

* The sample size of the study is 124 (for primiparous=62, multiparous=62).
* Frist, primiparous women who applied to the hospital for vaginal delivery will be divided into 2 arms as 31 experimental group and 31 control group.
* Second, multiparous women who applied to the hospital for vaginal delivery will be divided into 2 arms as 31 experimental group and 31 control group.

Data Collection Tools;

* Introductory Information Form,
* Visual Analog Scale for Pain,
* Wijma Birth Expectation/Experience Scale B version,
* Birth Satisfaction Scale

Application time:

* The neurolinguistic programming will be applied to the experimental group. NLP application will be done when the cervical opening is 4 cm, when the cervical opening is 5-6 cm, when the cervical opening is 7-8 cm.NLP application will be done three times in total. Each session will last 20 minutes
* No neurolinguistic programming will be applied to the control group.

Measurement time:

* Introductory Information Form will be completed by the woman when the cervical dilatation is 3-4 cm.
* VAS for pain will be measured before and immediately after the application when cervical dilatation is 4 cm; before and immediately after the application when cervical dilatation is 5-6 cm; before and immediately after the application when cervical dilatation is 7-8 cm; when cervical dilatation is 9-10 cm.
* Wijma Birth Expectation/Experience Scale B version and Birth Satisfaction Scale will be completed by the woman in the postnatal ward at approximately the second hour postpartum after the birth has taken place.
* The labour duration will be started for the mother who comes to the delivery room when the cervical opening is 4 cm and the total labour duration will be measured in minutes after the birth occurs.
* The control group will not be administered NLP only, but the measurements will be completed as in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women who give birth vaginally,
* whose birth takes place in the delivery room unit,
* who are 19 years of age or older and 35 years of age or younger,
* who are born at 37 and above gestational weeks,
* who give singleton birth,
* who do not have chronic diseases and any complications in this pregnancy and postpartum period

Exclusion Criteria:

* mothers who wish to leave the study voluntarily at any stage after being included in the study,
* who develop any health problems in themselves or their babies during the birth and postnatal period will be excluded from the scope.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 124 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-01-21 (Actual); Study Completion 2024-01-21 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for Pain | immediately before neuro linguistic programming application when the cervical opening was 4 cm, 5-6 cm, 7-8 cm
  Visual Analogue Scale for Pain; Scores between 0-10 are received. The difference in score indicates that the pain is aching.
Visual Analogue Scale for Pain | immediately after neurolinguistic programming application when the cervical opening was 4 cm, 5-6 cm, 7-8 cm
  Visual Analogue Scale for Pain; Scores between 0-10 are received. The difference in score indicates that the pain is aching.
Wijma Birth Anticipation/Experience Scale B version; | between approximately the second to sixth hours postpartum
  Wijma Birth Anticipation/Experience Scale B version; The minimum score from the scale is 0 and the maximum score is 165 points. If the total score obtained from the scale is below 66, it is considered mild, between 66 and 85, it is considered moderate, and above 85, it is considered severe fear of childbirth.
Birth Satisfaction Scale; | between approximately the second to sixth hours postpartum
  Birth Satisfaction Scale; The score that can be obtained from the scale is between 30-150 points. The change in the score obtained from the scale from birth increases.
Labour duration | the duration of labour will be calculated in minutes from the time the cervical opening begins until the fourth stage of labour
  Labour duration; time will be measured in minutes
Visual Analogue Scale for Pain | when the cervical opening was 9-10 cm
  Visual Analogue Scale for Pain; Scores between 0-10 are received. The difference in score indicates that the pain is aching.

CONTACTS AND LOCATIONS:
Locations (1):
- Şanlıurfa training and research hospital, Sanliurfa, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No